CLINICAL TRIAL: NCT02511587
Title: Comparison of Vaccination Routes: Subcutaneous Versus Intramuscular Application of FSME-Immun®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Univ. Prof. Dr. Ursula Wiedermann, Univ.-Prof. Dr. Ursula Wiedermann, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RV_FSME_1.2
Record Dates: First submitted 2015-07-23; First posted 2015-07-30 (Estimated); Results first posted 2018-05-18 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Vaccine Efficacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intra muscular application (Active Comparator): intra muscular application of FSME-Immune vaccination
  Interventions: Biological: FSME-Immune vaccination
- subcutaneous application (Experimental): subcutaneous application of FSME-Immune vaccination
  Interventions: Biological: FSME-Immune vaccination

INTERVENTIONS:
Biological: FSME-Immune vaccination — booster vaccination with FSME-Immune

SUMMARY:
FSME-Immun® is registered for application into the muscle. This study investigates if application under the skin leads to a comparable immune response.

DETAILED DESCRIPTION:
Tick-borne encephalitis (TBE) vaccine (FSME-Immun®) is registered for intra-muscular application. Due to medical reasons (e.g. anticoagulant therapy, adipositas) intra-muscular application is not always possible. The aim of this clinical trial is to investigate whether a comparably good immunogenicity can be achieved via the subcutaneous vaccination route. Thus humoral and cellular immune responses after intramuscular and subcutaneous TBE vaccination in healthy volunteers will be compared.

ELIGIBILITY:
Inclusion Criteria:

* completed primary TBE immunization + at least one booster immunization
* adults of both sexes between 18 and 60 years of age
* willingness to sign written informed consent form

Exclusion Criteria:

* age < 18 and > 60 years
* prior TBE infection
* pregnancy and breast feeding
* acute infection on day of inclusion (day 0), (body temperature > 37,9°C)
* concomitant medications: systemic cortisone therapy, chemotherapy, immunosuppressive therapy 4 weeks prior to or during study
* administration of other vaccines 4 weeks before/after day 0
* planned surgery within 2 weeks before/after TBE booster vaccination
* specific immunotherapy (Hypo-/Desensibilisation) 14 days before/after vaccination
* any contraindication to administration of FSME-Immun® vaccine according to manufacturer's instructions
* history of malignant disease within the last 5 years
* autoimmune diseases
* drug addictions
* plasma donors
* receipt of blood transfusions or immuno globulins within 3 month before study entry

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2012-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Wiedermann, MD, PhD, Principal Investigator — Medical University Vienna, ISPTM

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intra Muscular Application | Subcutaneous Application
Started | 58 | 58
Completed | 58 | 58
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intra Muscular Application | Subcutaneous Application | Total
Number analyzed (Participants) | 58 | 58 | 116
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 58 | 58 | 116
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 58
  Male | 29 | 29 | 58

OUTCOME MEASURES:

1. Primary Outcome: Humoral Immunity to TBE (Tick-borne Encephalitis) Vaccine
Description: GMT (geometric mean titers) of TBE Neutralisation test titers one month after booster vaccination
Time Frame: 1 month
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titers
Arm/Group | Intra Muscular Application | Subcutaneous Application
Number analyzed (Participants) | 58 | 58
Geometric mean titers | 574.8 [439 to 751] | 612.0 [483 to 775]

2. Secondary Outcome: Cellular Immune Responses - Cytokines
Description: cytokine production of antigen-specifically restimulated PMBC (peripheral blood mononuclear cells) is evaluated (Interleukin 2, Interleukin 10, Interferon gamma)
Time Frame: before (day 0) and 1 week after booster vaccination
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Intra Muscular Application | Subcutaneous Application
Number analyzed (Participants) | 58 | 58
pg/ml
  IFNg before vaccination | 2376 (2099) | 2199 (1781)
  IFNg one week post vacc | 3071 (2347) | 3387 (4375)
  IL-2 before vaccination | 81.8 (111.4) | 57.6 (66.1)
  IL-2 one week post vacc | 77.0 (97.8) | 56.5 (54.0)
  IL-10 before vaccination | 183.5 (219.8) | 192.8 (307.7)
  IL-10 one week post vacc | 210.6 (210.3) | 297.4 (343.3)

3. Secondary Outcome: TBE Titer Profile
Description: TBE specific neutralizing antibody titer profiles (geometric mean titers, GMT)
Time Frame: before (day 0) and 1week, 1 month, 6 months after booster vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titers
Arm/Group | Intra Muscular Application | Subcutaneous Application
Number analyzed (Participants) | 58 | 58
Geometric mean titers
  GMT at d0 | 249.9 [185.3 to 337.1] | 208.8 [159.2 to 273.8]
  GMT after 1 week | 360.9 [278.8 to 467.2] | 317.2 [245.1 to 410.6]
  GMT after one month | 574.8 [439.5 to 751.6] | 612.0 [483 to 775.4]
  GMT after 6 month | 420.1 [318.5 to 554.2] | 380.5 [293.5 to 493.5]

ADVERSE EVENTS:
Arm/Group | Intra Muscular Application | Subcutaneous Application
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/58
Other Adverse Events (participants affected / at risk) | 0/58 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes